CLINICAL TRIAL: NCT02030223
Title: The Analgesic Efficacy of the Ultrasound Guided Transversus Abdominis Plane Block After Inguinal Hernia Repair With a Mesh.
Brief Title: Transversus Abdominis Plane Block and Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papacharalampous Panagiota (Other)
Responsible Party: Sponsor-Investigator, Papacharalampous Panagiota, Anesthesiologist, Aretaieion University Hospital
Organization: Aretaieion University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAM-2345-1786
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Inguinal Hernia; Abdominal Wall Muscles; Regional Anesthesia; Postoperative Pain
Keywords: transversus abdominis plane block; inguinal hernia repair; acute postoperative pain; neuropathic pain
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transversus abdominis plane block with 20 ml ropivacaine 0,75% (Active Comparator): Transversus abdominis plane block with 20 ml ropivacaine 0,75%
  Interventions: Procedure: Transversus abdominis plane block
- Transversus abdominis plane block with 20 ml saline (Placebo Comparator): Transversus abdominis plane block with 20 ml saline
  Interventions: Procedure: Transversus abdominis plane block

INTERVENTIONS:
Procedure: Transversus abdominis plane block — ultrasound guided transversus abdominis plane block

SUMMARY:
This prospective, randomized, double blinded, placebo-controlled study is designed to evaluate the postoperative analgesic efficacy of the ultrasound-guided transversus abdominis plane block with ropivacaine 0,75 %, in patients undergoing unilateral inguinal hernia repair with a mesh under general anaesthesia, and how the efficiency of early postoperative analgesia achieved correlates with the risk of developing a chronic pain state, a not uncommon condition after this type of surgery.

ELIGIBILITY:
Inclusion Criteria:

ASA I-III patients undergoing inguinal hernia repair with a mesh

age between 18 and 75 years old

ability to read and write greek

-

Exclusion Criteria:

* Inability to consent to the study
* BMI >40kg/m2
* Skin infection at the puncture site
* Contraindication to mono-amide local anaesthetics, paracetamol, NSAID's (parecoxib)
* Preoperative use of opioids or NSAID's for chronic pain conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pain scores at rest and with movement using the numerical rating scale (NRS) | 3, 6 and 24 hours postoperatively

SECONDARY OUTCOMES:
Incidence of chronic pain | 6 months after surgery

OTHER OUTCOMES:
Morphine consumption (mg) | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Erifyli Argyra, MD, PhD, Study Chair — Aretaieion University Hospital; Kassiani Theodoraki, MD, PhD, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Greece

REFERENCES:
- [Result] Milone M, Di Minno MN, Musella M, Maietta P, Salvatore G, Iacovazzo C, Milone F. Outpatient inguinal hernia repair under local anaesthesia: feasibility and efficacy of ultrasound-guided transversus abdominis plane block. Hernia. 2013 Dec;17(6):749-55. doi: 10.1007/s10029-012-1022-2. Epub 2012 Nov 16. PMID 23160979
- [Result] Petersen PL, Mathiesen O, Stjernholm P, Kristiansen VB, Torup H, Hansen EG, Mitchell AU, Moeller A, Rosenberg J, Dahl JB. The effect of transversus abdominis plane block or local anaesthetic infiltration in inguinal hernia repair: a randomised clinical trial. Eur J Anaesthesiol. 2013 Jul;30(7):415-21. doi: 10.1097/EJA.0b013e32835fc86f. PMID 23549122
- See also: THE JOURNAL OF THE NEW YORK SCHOOL OF REGIONAL ANESTHESIA — http://WWW.NYSORA.COM